CLINICAL TRIAL: NCT07045805
Title: Phase II Study of Iparomlimab and Tuvonralimab Combined With Paclitaxel and Bevacizumab for the Treatment of Advanced Gastric or Gastroesophageal Junction Adenocarcinoma That Failed First-Line Treatment With PD-(L)1 Inhibitor Combined With Chemotherapy
Brief Title: Phase II Study of QL1706 Combined With Paclitaxel and Bevacizumab for Second-Line Immune Rechallenge in Gastric Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Jia Wei, MD, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QL-GasC-QIBA-1002
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Gastric Cancer (GC)
MeSH Terms: conditions — Stomach Neoplasms | interventions — Paclitaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QL1706 combined with paclitaxel and bevacizumab (Experimental): QL1706 7.5 or 5 mgmg/kg combined with paclitaxel 150 mg/m2 and bevacizumab 7.5mg/kg, d1, Q3W
  Interventions: Drug: QL1706 combined with paclitaxel and bevacizumab

INTERVENTIONS:
Drug: QL1706 combined with paclitaxel and bevacizumab — Phase 1:
  Plan to enroll 6 subjects to receive QL1706 7.5 mg/kg, paclitaxel 150 mg/m², and bevacizumab 7.5 mg/kg, d1, Q3W. Subjects will undergo a 3-week Dose-Limiting Toxicity (DLT) evaluation period.
  If ≥2 DLTs occur among the 6 subjects, QL1706 5 mg/kg will be selected as the Recommended Phase 2 Dose (RP2D) for Phase 2.
  Otherwise, QL1706 7.5 mg/kg will be the RP2D for Phase 2.
  Phase 2:
  Plan to enroll 54-60 subjects. Starting from Cycle 1, QL1706 will be administered intravenously at the RP2D determined in Phase 1. Subjects will receive:
  QL1706 (RP2D) Paclitaxel 150 mg/m² Bevacizumab 7.5 mg/kg All agents administered on day 1 of each Q3W cycle. Treatment Duration for All Subjects: Continues until disease progression, intolerable toxicity, withdrawal of informed consent, death, or initiation of new antitumor therapy-whichever occurs first.

SUMMARY:
The study aims to evaluate the efficacy and safety of the QL1706 combination with paclitaxel and bevacizumab in patients with gastric adenocarcinoma and gastroesophageal junction adenocarcinoma who have failed first-line standard therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent and voluntarily enrolled in the study.
2. Aged 18-75 years, regardless of gender.
3. Histologically or cytologically confirmed unresectable or metastatic gastric or gastroesophageal junction adenocarcinoma.
4. Documented failure after ≥3 cycles of prior first-line PD-(L)1 inhibitor combined with fluorouracil-based or platinum-based chemotherapy.

   *Note: Disease recurrence/progression ≤6 months after completing (neo)adjuvant systemic therapy qualifies as first-line treatment.*
5. HER2-negative status (IHC 0/1+ or IHC 2+/FISH-negative).
6. ECOG Performance Status 0-1.
7. ≥1 measurable lesion per RECIST v1.1. Previously irradiated lesions cannot be target lesions unless: the irradiated lesion is the sole measurable lesion and documented progression in the irradiated lesion by imaging
8. Life expectancy ≥3 months.
9. Adequate organ function:

   1. Hematology (no blood products/growth factors within 14 days prior):

      * Absolute neutrophil count ≥1.0×10⁹/L
      * Platelets ≥75×10⁹/L
      * Hemoglobin ≥90 g/L
   2. Biochemistry:

      * Total bilirubin ≤1.5×ULN
      * ALT/AST ≤2.5×ULN (≤5×ULN if liver metastases)
      * Serum creatinine ≤1.5×ULN or creatinine clearance ≥50 mL/min
   3. Coagulation:

      * INR ≤1.5×ULN
      * aPTT ≤1.5×ULN
10. Reproductive requirements:

    * Females of childbearing potential: Negative serum/urine pregnancy test within 72h prior to dosing; use effective contraception (IUD/oral contraceptives/condoms) during treatment and ≥120 days post-last dose.
    * Males with fertile partners: Surgical sterilization or agreement to use effective contraception during treatment and ≥120 days post-last dose.
11. Willingness to comply with protocol-specified follow-up procedures.

Exclusion Criteria:

1. Histopathological or cytological examination confirms the presence of other pathological components, such as squamous cell carcinoma, undifferentiated carcinoma, neuroendocrine carcinoma, etc.
2. Previous systemic treatment targeting VEGF or the anti-VEGFR signaling pathway.
3. Previous treatment with PD-1/CTLA-4 dual immunotherapy.
4. Previous systemic or local treatment with paclitaxel-based drugs.
5. Received the last anti-tumor therapy within 5 half-lives (whichever is shorter) prior to the first dose, including chemotherapy, immunotherapy, targeted therapy (within 2 weeks prior to the first dose for small molecule targeted therapy), biological therapy, etc.; Palliative local therapy for non-target lesions within 2 weeks prior to the first dose; Received systemic non-specific immunomodulatory therapy (e.g., interleukin, interferon, thymosin) within 2 weeks prior to the first dose.
6. History of Grade 3 or higher irAEs (excluding endocrine system-related irAEs) caused by PD-1/PD-L1 inhibitors.
7. Permanent discontinuation of previous treatment due to irAEs.
8. Has not adequately recovered (i.e., ≤ Grade 1 or returned to baseline, excluding fatigue or alopecia) from toxicities and/or complications caused by any prior intervention prior to starting treatment.
9. Presence of clinically symptomatic pleural effusion, pericardial effusion, or ascites requiring frequent drainage (≥1 time/month).
10. Known active or untreated brain metastases, leptomeningeal metastases, spinal cord compression, or leptomeningeal disease. However, subjects with measurable disease outside the central nervous system who meet the following criteria may be enrolled: asymptomatic after treatment, radiologically stable for at least 4 weeks prior to initiation of study treatment (e.g., no new or enlarging brain metastases), and off systemic glucocorticoids and anticonvulsants for at least 2 weeks.
11. History of gastrointestinal perforation, gastrointestinal fistula, or intra-abdominal abscess within 6 months prior to the first dose.
12. History of bowel obstruction and/or clinical signs or symptoms of gastrointestinal obstruction within 6 months prior to the first dose, including incomplete obstruction related to the underlying disease or requiring routine parenteral hydration, parenteral nutrition, or tube feeding.
13. Significant clinically significant bleeding symptoms or definite bleeding tendency within 6 months prior to the first dose, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, or vasculitis, etc., excluding asymptomatic occult blood-positive stool.
14. Tumor invasion of major blood vessels, or investigator judgment based on imaging that tumor invasion of major blood vessels is highly likely during the future study period, potentially leading to fatal hemorrhage.
15. Arterial or venous thromboembolic events within 6 months prior to the first dose, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism, etc. (superficial venous thrombosis is allowed).
16. Major surgery (as determined by the investigator), open biopsy, or significant trauma within 28 days prior to the first dose; or planned elective major surgery during the study period.
17. Urinalysis indicates urine protein ≥ ++ and confirmed 24-hour urine protein > 1.0 g.
18. Hypertension that cannot be adequately controlled with antihypertensive medication (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg); History of hypertensive crisis or hypertensive encephalopathy.
19. Serious infection (CTCAE > Grade 2) within 4 weeks prior to the first study drug dose, such as severe pneumonia requiring hospitalization, bacteremia, or complicated infections; Active pulmonary inflammation indicated by baseline chest imaging; Signs/symptoms of infection within 14 days prior to the first dose or requiring oral/intravenous antibiotics (excluding prophylactic antibiotic use).
20. Any active autoimmune disease or history of autoimmune disease, including but not limited to: interstitial pneumonia, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism (may be considered if controlled with hormone replacement therapy); Subjects with psoriasis or childhood asthma/allergies in complete remission without adult intervention may be considered; patients requiring medical intervention with bronchodilators are excluded.
21. History of immunodeficiency, including positive HIV test, or other acquired/congenital immunodeficiency diseases, or history of organ transplantation or allogeneic bone marrow transplantation.
22. Poorly controlled cardiac clinical symptoms or diseases, including but not limited to: (1) NYHA Class II or higher heart failure, (2) unstable angina, (3) myocardial infarction within 1 year, (4) clinically significant supraventricular or ventricular arrhythmias uncontrolled without or despite clinical intervention; (5) QTc > 450ms (male); QTc > 470ms (female).
23. Active tuberculosis infection identified by history or CT scan, or history of active tuberculosis infection within 1 year prior to enrollment, or history of active tuberculosis infection more than 1 year ago without formal treatment.
24. Active hepatitis (Hepatitis B reference: HBsAg positive and HBV DNA ≥2000 IU/mL; Hepatitis C reference: HCV antibody positive and HCV RNA > upper limit of normal).
25. Diagnosed with other malignancies within 5 years prior to the first study drug dose, except for malignancies with low risk of metastasis or death (5-year survival rate > 90%), such as adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix, etc., who may be considered for enrollment.
26. Received live attenuated vaccines within 4 weeks prior to the first study drug dose; If enrolled, subjects must not receive live vaccines during the study or within 120 days after the last dose of eplonolimab tovorilimab.
27. Known allergy or intolerance to any study drug(s) and/or any excipients.
28. Pregnant or lactating women.
29. Currently participating in another clinical study, unless it is an observational, non-interventional study or in the follow-up period of an interventional study.
30. Other factors that, in the investigator's judgment, may lead to premature termination from the study, such as other severe diseases (including psychiatric disorders) requiring combined treatment, alcoholism, drug abuse, familial or social factors, or any other factors affecting subject safety or compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-07-25 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
PFS | up to 7 months
  The time from the initiation of the first dose to the occurrence of disease progression or death, whichever comes first.
Dose-limiting toxicity | Within Cycle 1 (21 days)

SECONDARY OUTCOMES:
OS | up to 13 months
  The time interval between the start date of study drug and the date of death (any cause)
DoR | up to 6 months
  monitor the length of time patients experience a reduction in tumor size or stabilization of disease following the treatment
ORR | up to 7 months
  the proportion of subjects achieving complete response (CR) or partial response (PR)
AE | the first dose until 90 days after the last dose of QL1706 or 30 days after the last dose of other study drugs, whichever comes later.
  Number and percentage of participants with Adverse Events(any grade)

IPD SHARING:
Plan to Share IPD: No